CLINICAL TRIAL: NCT04687904
Title: Mindfulness Meditation for Epilepsy: Effect of Mindfulness Meditation Practice on Quality of Life and EEG Activity in Refractory Epilepsy
Brief Title: Mindfulness Meditation for Epilepsy
Acronym: MIME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Collaborators: Laboratoire Traitement du Signal et de l'Image, INSERM UMR1099 Rennes (Unknown); Centre Hospitalier Guillaume Régnier, RENNES (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35RC20_8848; 2020-A02336-33 (Other: Id-RCB)
Record Dates: First submitted 2020-12-18; First posted 2020-12-29 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Epilepsy
Keywords: Mindfulness meditation
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic education group (Active Comparator): The psychologist associated with the project takes care of the patient to receive a 1.5 hour therapeutic education interview ("control" group).
  Interventions: Behavioral: Therapeutic education
- Mindfulness meditation group (Experimental): The psychologist associated with the project takes care of the patient to receive training in mindfulness meditation twice (1.5 hours) ("active" group)
  Interventions: Behavioral: Mindfulness meditation training

INTERVENTIONS:
Behavioral: Mindfulness meditation training — Patients will be able to benefit from mindfulness meditation training at the rate of 1h30 in the morning and 1h30 in the afternoon. During this training, patients will be invited to share with the psychologist their vision of mindfulness meditation and their expectations of this practice. The psychologist will then introduce what mindfulness is and how the sessions will take place. Several sessions guided by the psychologist will then be offered to the patient (body scan, focused attention, mindfulness movements...).
  Arms: Mindfulness meditation group
Behavioral: Therapeutic education — Patients will benefit from a 2-hour interview which will be conducted by the psychologist associated with the project.
  The aim of this interview is to help patients better understand their disease in order to adopt the right behaviors on a daily basis. This session will inform patients about their disease, its origins, its treatment, the difficulties it causes and the means to remedy it. The objective of this session is to better understand and manage epilepsy and to enable patients to take an active part in the process of care and management of the disease.
  No specific instructions will be given at the end of this interview.
  Arms: Therapeutic education group

SUMMARY:
In one-third of epileptic patients treated in France, seizures persist despite drug treatment. These so-called "refractory" epilepsies are among the most severe. Only a minority of patients with refractory epilepsy can undergo surgery. The other options available are based on brain or vagus nerve stimulation interventions which clinical effectiveness is still being studied. Alternative therapies are needed both to decrease the frequency of patients' seizures and to improve their quality of life.

The practice of mindfulness meditation has recently been included in the recommendations of the International League Against Epilepsy in order to alleviate anxiety or depression comorbid symptoms.

This study falls within this framework by targeting two aspects of the pathology.

DETAILED DESCRIPTION:
Through the development of standardized protocols, mindfulness meditation has been introduced as a complementary treatment to prevent the relapse of depression, and to reduce stress and improve well-being in many chronic conditions.

Epilepsy, which results from the activity of hyperexcitable circuits, is also associated with a disorganization of the physiological brain networks. Studies in cognitive neuroscience in healthy subjects suggest that meditation induces lasting changes in the physiological networks of attention and default mode and could potentially compensate for dysfunctions of these networks in epileptic patients.

ELIGIBILITY:
Inclusion Criteria:

* For patients :

  * Patients over 16 years of age;
  * Epilepsy refractory to drug treatment according to the consensus criteria of the International League Against Epilepsy ;
  * Affiliated with a health insurance plan;
  * Free, informed and written consent signed by the patient, and parents for patients under the age of 18.
* For healthy subjects :

  * Healthy subjects 16 years of age and older;
  * Affiliated with a health insurance plan;
  * Free, informed and written consent signed by the volunteer, or parents, for volunteers under the age of 18.

Exclusion Criteria:

* For patients :

  * Alcohol Addiction Disorders (assessed by the Mini-International Neuropsychiatric Interview (MINI) scale) ;
  * Patients with psychogenic crises;
  * Treatment with antidepressants;
  * Simultaneous participation in other research that may interfere with the protocol;
  * Persons of legal age subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty.
* For healthy subjects :

  * Psychiatric pathology and/or alcohol addiction disorders (evaluated by the MINI scale) ;
  * Simultaneous participation in other research that may interfere with the protocol;
  * Persons of legal age subject to legal protection (protection of justice, guardianship, trusteeship), persons deprived of liberty.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
Short Form Quality of Life Questionnaire (SF36) score at 3 months | At inclusion and at 3 months
  Change in the score on the Short Form Quality of Life Questionnaire (SF36) assessed before the intervention and at 3 months.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

SECONDARY OUTCOMES:
Short Form Quality of Life Questionnaire (SF36) score at 1 months | At inclusion and at 1 month
  Change in the score on the Short Form Quality of Life Questionnaire (SF36) assessed before the intervention and at 1 month.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Depressive symptoms assessed on the Montgomery-Åsberg Depression Rating Scale (MADRS) at 1 month | At inclusion and at 1 month
  MADRS score is evaluated before the intervention and at 1 month. Montgomery Äsberg Depression Rating Scale (MADRS): is a scale of depression (diagnosis + follow-up evolution, therapeutic response criteria). It consists of 10 items rated from 0 to 6 from a semi-structured interview, to obtain a total depression score of 0 to 60 (0 no depression, 60 maximum depression intensity). Items evaluate: apparent sadness, expressed sadness, inner tension, reduced sleep, reduced appetite, difficulty concentrating, weariness, inability to feel, pessimistic thoughts, thoughts of suicide ;
Depressive symptoms assessed on the Evolution of MADRS score at 3 months | At inclusion and at 3 months
  MADRS score is evaluated before the intervention and at 3 months. Montgomery Äsberg Depression Rating Scale (MADRS): is a scale of depression (diagnosis + follow-up evolution, therapeutic response criteria). It consists of 10 items rated from 0 to 6 from a semi-structured interview, to obtain a total depression score of 0 to 60 (0 no depression, 60 maximum depression intensity). Items evaluate: apparent sadness, expressed sadness, inner tension, reduced sleep, reduced appetite, difficulty concentrating, weariness, inability to feel, pessimistic thoughts, thoughts of suicide ;
Depressive symptoms assessed on the Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) at 1 month | At inclusion and at 1 month
  NDDI-E score is evaluated before the intervention and at 1 month. Depression scale score 0 to 24
Depressive symptoms assessed on the Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) at 3 months | At inclusion and at 3 months
  NDDI-E score is evaluated before the intervention and at 3 months. Depression scale score 0 to 24
Anxiety symptoms assessed on the State-Trait Anxiety Inventory scale (STAI) at 1 month. | At admission and at 1 month
  Scores on the State-Trait Anxiety Inventory scale (STAI A and B) evaluated before the intervention and at 1 month.
  STAI (State Trait Anxiety Inventory) form A and B: is an anxiety scale. The first part concerns state anxiety and consists of a self-questionnaire of 20 items, the subject having to score on a 4-point Likert scale (not at all, little, moderately, much) his current anxiety level. The second part concerns trait anxiety and consists of a self-questionnaire of 20 items, the subject having to score on a 4-point Likert scale (almost never, sometimes, often, almost always) his level of background anxiety. Two scores varying between 10 (minimum anxiety) and 40 (maximum anxiety) are therefore obtained;
Anxiety symptoms assessed on the State-Trait Anxiety Inventory scale (STAI) at 3 months. | At inclusion and at 3 months
  Scores on the State-Trait Anxiety Inventory scale (STAI-Y A and B) evaluated before the intervention and at 3 months.
  STAI (State Trait Anxiety Inventory) form A and B: is an anxiety scale. The first part concerns state anxiety and consists of a self-questionnaire of 20 items, the subject having to score on a 4-point Likert scale (not at all, little, moderately, much) his current anxiety level. The second part concerns trait anxiety and consists of a self-questionnaire of 20 items, the subject having to score on a 4-point Likert scale (almost never, sometimes, often, almost always) his level of background anxiety. Two scores varying between 10 (minimum anxiety) and 40 (maximum anxiety) are therefore obtained;
Anxiety symptoms assessed on the General Anxiety Disorder 7 scale (GAD-7) at 1 month. | At admission and at 1 month
  Scores on GAD-7 scale evaluated before the intervention and at 1 month. Generalised anxiety disorder score (GAD-7) scale. Score 0-21, with a higher score associated with greater anxiety symptoms. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. GAD-7 score at baseline will be controlled for.
Anxiety symptoms assessed on the General Anxiety Disorder 7 scale (GAD-7) at 1 month. | At admission and at 3 months
  Scores on GAD-7 scale evaluated before the intervention and at 3 months. Generalised anxiety disorder score (GAD-7) scale. Score 0-21, with a higher score associated with greater anxiety symptoms. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. GAD-7 score at baseline will be controlled for.
Seizure frequency at 1 month | At 1 month
  Seizure frequency: self-assessed by the patient and those around him/her using a seizure diary.
Seizure frequency at 3 month | At 3 month
  Seizure frequency: self-assessed by the patient and those around him/her using a seizure diary.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle MERLET, PhD, Study Chair — LTSI - INSERM UMR 1099
Locations (1):
- Centre Hospitalier Universitaire, Rennes, France